CLINICAL TRIAL: NCT06834334
Title: Clinical Effectiveness of Advanced Hybrid Closed-loop Systems (AHCL) for Achieving Time in Tight Range (TiTR) of Interstitial Glucose Among Adult Type 1 Diabetes (T1D) Patients
Brief Title: Clinical Effectiveness of Advanced Hybrid Closed-loop Systems for Achieving Time in Tight Range Among T1D Patients
Acronym: TightT1
Status: Recruiting | Type: Observational
Sponsor: Castilla-La Mancha Health Service (Other)
Collaborators: Servicio Extremeño de Salud (Spain) (Unknown); Hospital Universitari Mutua Terrassa (Unknown)
Responsible Party: Sponsor
Other Study IDs: C-790
Record Dates: First submitted 2025-02-07; First posted 2025-02-19 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Type 1 Diabetes (T1D)
Keywords: Type 1 diabetes; Advanced hybrid closed-loop; Time in tight range; artificial pancreas; Control-IQ; SmartGuard; CamAPS
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- MM780G: Patients with type 1 diabetes treated with Medtronic Minimed 780G hybrid closed-loop systems
  Interventions: Device: MM780G
- TTSX2: Patients with type 1 diabetes treated with Tandem T Slim X2 hybrid closed-loop system
  Interventions: Device: TTSX2
- CamAPS: Patients with type 1 diabetes treated with CamAPS hybrid closed-loop system
  Interventions: Device: CamAPS

INTERVENTIONS:
Device: MM780G — SmartGuard in Medtronic Minimed 780G advaced hybrid closed-loop
  Other Names: Medtronic Minimed 780G
  Groups: MM780G
Device: TTSX2 — Control-IQ in Tandem T Slim X2 advanced hybrid closed-loop
  Other Names: Tandem T Slim X2
  Groups: TTSX2
Device: CamAPS — CamAPS Fx in Ypsopump advanced hybrid closed-loop
  Other Names: CamAPS Fx
  Groups: CamAPS

SUMMARY:
Diabetes is a chronic disease with a relevant public health burden. Maintaining blood glucose levels as close to normal as possible is essential to avoid the associated microvascular and macrovascular complications. Therefore, the key to prevent and/or reduce the development of these chronic complications lies in an adequate and strict glycemic control.

This study consist of a cross-sectional observational study among adult patients with type 1 diabetes (T1D). The main objective is to analyze the effect on time in tight range (TiTR, 70-140 mg/dL) of interstitial glucose between three different advanced hybrid closed-loop (AHCL) systems.

DETAILED DESCRIPTION:
Diabetes is a chronic disease with a relevant public health burden. Type 1 diabetes (T1D) is characterized by the autoimmune destruction of insulin-producing pancreatic beta cells, which requires the administration of exogenous insulin for its treatment. Maintaining blood glucose levels as close to normal as possible is essential to avoid the associated microvascular and macrovascular complications that affect quality of life, as well as morbidity and mortality due to the deleterious long-term effects of suboptimal control. Therefore, the key to prevent and/or reduce the development of these complications lies in adequate and strict glycemic control.

The use of advanced hybrid closed-loop (AHCL) systems in patients with T1D is associated with improved glycemic control and quality of life in both controlled clinical trials and real-life studies. Since 2021, AHCL systems are considered the standard of care, ahead of traditional MDI.

There are three main types of AHCL systems marketed in Spain: SmartGuard in Medtronic Minimed 780G (MM780G), Control-IQ in Tandem T Slim X2 (TTSX2) and CamAPS in Ypsopump (CamAPS).

All three systems have been shown indepently to significantly improve glycaemic control in people with DM1 as expressed by the classic control targets of the International Time in Range Consensus (percentage of interstitial glucose time in range 70-180 mg/dL >70%). So much so that it has been suggested to further intensify the possible glucose targets in patients treated with AHCL systems to a time in tight range (TITR) of interstitial glucose (70-140 mg/dL) >50%.

However, there is little information on the benefits and safety of using tighter control targets. Furthermore, there is no evidence about comparing the clinical benefit differences between these three types of technology.

The main objective is to analyze the effect on time in tight range (TiTR, 70-140 mg/dL) of interstitial glucose between three different advanced hybrid closed-loop (AHCL) systems among adult people with T1D.

This is multicenter (3 centers) cross-sectional observational clinical study (non-randomized). The target population will be adult T1D patients treated with any of the aforementioned AHCL systems followed in any of the three participant centers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 diabetes.
* Age greater than or equal to 18 years.
* Treated with advanced hybrid closed-loop systems (AHCL) for at least 3 months
* Actived continuous glucose monitoring data in the last 14 days.

Exclusion Criteria:

* Other types of diabetes.
* Receiving treatment with insulin regimens other than AHCL.
* Having received AHCL treatment for less than 3 months in a row prior to inclusion in the study with the same system.
* No data on use of the AHCL system during the previous 14 days.
* Severe or uncontrolled psychiatric disorder.
* Pregnancy or end of pregnancy less than 3 months ago or preparation for pregnancy.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with type 1 diabetes treated with AHCL attended in any of the three centers.
Sampling Method: Non-Probability Sample
Enrollment: 189 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
TiTR | Retrospective data from the last 14 days after study entry
  Percentage differences in time in tight range (TiTR, 70-140 mg/dL) of interstitial glucose.

SECONDARY OUTCOMES:
TIR | Retrospective data from the last 14 days after study entry
  Percentage differences in time in range (TIR, 70-180 mg/dL) of interstitial glucose.
TAR1 | Retrospective data from the last 14 days after study entry
  Percentage differences in time above range 1 (180-250 mg/dL) of interstitial glucose.
TAR2 | Retrospective data from the last 14 days after study entry
  Percentage differences in time above range 2 (>250 mg/dL) of interstitial glucose.
TBR1 | Retrospective data from the last 14 days after study entry
  Percentage differences in time bellow range 1 (<70 mg/dL) of interstitial glucose.
TBR2 | Retrospective data from the last 14 days after study entry
  Percentage differences in time bellow range 2 (<55 mg/dL) of interstitial glucose.
HbA1C | Retrospective data from the last 3 months after study entry
  Differences in HbA1C values (%)
AHCL use | Retrospective data from the last 14 days after study entry
  Percentage differences in time of use of the AHCL system (%)
Insulin use | Retrospective data from the last 14 days after study entry
  Daily dose of insulin use in AHCL system (UI/day)
Coefficient of variation | Retrospective data from the last 14 days after study entry
  Percentage differences in the coefficient of variation of interstitial glucose (%)
Quality-of-life questionnaire designed for diabetes mellitus (EsDQOL) | Retrospective quality-of-life during the last 3 months
  Assessing the perceived quality of life according to the EsDQOL questionnaire (with values between 46 and a maximum of 230, the higher the score the poorer the satisfaction with ACHL treatment).
Hypoglycemia Fear Survey (HFS questionnaire) | Retrospective fear to hypoglycemia during the last 3 months
  Assessing the fear of hypoglycemia according to the HFS questionnaire (with values between 24 points and a maximum of 120 points, the higher the score the higher the fear of hypoglycemia).
Clarke's questionnaire | Retrospective hypoglycemia awareness during the last 3 months
  Assessing the awareness of hypoglycemia according to Clarke's questionnaire (with values between 0 and 8 points, a score equal or greater than four indicates hypoglycemia unawareness).

OTHER OUTCOMES:
Differences in the Percetage of patients fullfilling the International Consensus of Time in Range | Retrospective data from the last 14 days after study entry
  Differences in the Percetage of patients fullfilling the International Consensus of Time in Range (TAR2 <5%, TAR1 <25%, TIR >70%, TBR1 <4%, TBR2 <1%, CV>36%).

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Moreno Fernandez, PhD, Principal Investigator — Castilla-La Mancha Health Public Service
Locations (3):
- Spain (3):
  - Badajoz University Hospital, Badajoz, Badajoz
  - Hospital Universitario Mutua de Tarrasa, Terrassa, Barcelona
  - Ciudad Real General University Hospital, Ciudad Real, Ciudad Real

IPD SHARING:
Plan to Share IPD: Undecided
Under request and after consideration from all investigators.

REFERENCES:
- [Background] American Diabetes Association Professional Practice Committee. 7. Diabetes Technology: Standards of Care in Diabetes-2024. Diabetes Care. 2024 Jan 1;47(Suppl 1):S126-S144. doi: 10.2337/dc24-S007. PMID 38078575
- [Background] Di Molfetta S, Di Gioia L, Caruso I, Cignarelli A, Green SC, Natale P, Strippoli GFM, Sorice GP, Perrini S, Natalicchio A, Laviola L, Giorgino F. Efficacy and Safety of Different Hybrid Closed Loop Systems for Automated Insulin Delivery in People With Type 1 Diabetes: A Systematic Review and Network Meta-Analysis. Diabetes Metab Res Rev. 2024 Sep;40(6):e3842. doi: 10.1002/dmrr.3842. PMID 39298688
- [Background] Beck RW, Kanapka LG, Breton MD, Brown SA, Wadwa RP, Buckingham BA, Kollman C, Kovatchev B. A Meta-Analysis of Randomized Trial Outcomes for the t:slim X2 Insulin Pump with Control-IQ Technology in Youth and Adults from Age 2 to 72. Diabetes Technol Ther. 2023 May;25(5):329-342. doi: 10.1089/dia.2022.0558. Epub 2023 Apr 12. PMID 37067353
- [Background] Castaneda J, Arrieta A, van den Heuvel T, Battelino T, Cohen O. Time in Tight Glucose Range in Type 1 Diabetes: Predictive Factors and Achievable Targets in Real-World Users of the MiniMed 780G System. Diabetes Care. 2024 May 1;47(5):790-797. doi: 10.2337/dc23-1581. PMID 38113453
- [Background] Beck RW, Raghinaru D, Calhoun P, Bergenstal RM. A Comparison of Continuous Glucose Monitoring-Measured Time-in-Range 70-180 mg/dL Versus Time-in-Tight-Range 70-140 mg/dL. Diabetes Technol Ther. 2024 Mar;26(3):151-155. doi: 10.1089/dia.2023.0380. Epub 2023 Oct 13. PMID 37870460
- [Background] Beato-Vibora PI, Chico A, Moreno-Fernandez J, Bellido-Castaneda V, Nattero-Chavez L, Picon-Cesar MJ, Martinez-Brocca MA, Gimenez-Alvarez M, Aguilera-Hurtado E, Climent-Biescas E, Azriel-Mir S, Rebollo-Roman A, Yoldi-Vergara C, Pazos-Couselo M, Alonso-Carril N, Quiros C. A Multicenter Prospective Evaluation of the Benefits of Two Advanced Hybrid Closed-Loop Systems in Glucose Control and Patient-Reported Outcomes in a Real-world Setting. Diabetes Care. 2024 Feb 1;47(2):216-224. doi: 10.2337/dc23-1355. PMID 37948469